CLINICAL TRIAL: NCT00109421
Title: PROJECT ÒRÉ: An Innovative Friendship Based HIV/STI Intervention for High Risk African American Females
Brief Title: Friendship Based HIV/STI (Sexually Transmitted Infections) Intervention for African American Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATN 034
Record Dates: First submitted 2005-04-27; First posted 2005-04-28 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: Sexual Behavior; Sexually Transmitted Diseases; HIV Infections
Keywords: adolescent; female; community-based; social network; HIV/STI intervention; High HIV-risk African American adolescent females
MeSH Terms: conditions — Sexual Behavior; Sexually Transmitted Diseases; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental arm (Experimental): In the experimental condition, the intervention group will receive the half-day Project ÒRÉ intervention. All participants will complete pre-, post- and 3-month follow-up self-administered questionnaires. A subset of groups will participate in a process evaluation focus group immediately following the program.
  Interventions: Behavioral: Project ÒRÉ
- Attention control group (No Intervention): The attention control group will receive a standard health promotion control program which has been used previously with similar populations. All participants will complete pre-, post- and 3-month follow-up self-administered questionnaires.

INTERVENTIONS:
Behavioral: Project ÒRÉ — Community-based adolescent social network HIV/STI intervention tailored to African American culture
  Other Names: ÒRÉ
  Arms: Experimental arm

SUMMARY:
The Project ÒRÉ intervention is a half-day community-based HIV/STI intervention program for friendship groups of adolescents that is tailored to African American culture. The four participating community sites will be assigned to either the Project ÒRÉ intervention or a standard health promotion program. Sexually experienced African American adolescent females will recruit members of their friendship group for the five-hour program. All participants will complete questionnaires before and immediately following the programs and another one 3 months later. Immediately following the program some of the Project ÒRÉ groups will also participate in a focus group to provide feedback about the program.

DETAILED DESCRIPTION:
A group-randomized controlled design to test the efficacy of the Project ÒRÉ intervention, a community-based adolescent social network HIV/STI intervention tailored to African American culture. Four community based organization sites (CBOs) will be randomly assigned to an experimental or attention control condition. In both conditions, sexually experienced African American adolescent females will recruit members of their friendship group for the five-hour program. In the experimental condition, the intervention group will receive the half-day Project ÒRÉ intervention. The attention control group will receive a standard health promotion control program which has been used previously with similar populations. All participants will complete pre-, post- and 3-month follow-up self-administered questionnaires. In the experimental condition, a subset of groups will participate in a process evaluation focus group immediately following the program.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between the ages of 14-18
* Self-identifies as African American
* Sexually experienced
* Willing to participate in a single five-hour workshop and a one-hour follow-up session
* Willing to nominate 2-5 close female friends ages 14-21 to participate in the study with her
* Lives in the experimental intervention community
* Ability to obtain permission from parent or legal guardian and assent from minors or consent from those above age of majority

Exclusion Criteria:

* Individual reports predominantly same gender sexual behavior
* Recent homelessness
* Visibly distraught or unstable (i.e. suicidal, manic, exhibiting violent behavior, etc.)
* Intoxicated or under the influence of psychoactive agents

Ages: 14 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 420 (Actual)
Dates: Start 2004-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Conduct elicitation research in the study community | 18 Months
  To conduct elicitation research in the study community to: assess the applicability of the existing Project ÒRÉ intervention modules, modify the intervention for the specific populations that are targeted in the current study, and incorporate local data in the production of three brief videos involving youth in the study community

SECONDARY OUTCOMES:
Test the efficacy of the intervention | 18 Months
  To use a group-randomized controlled design to conduct a test of the efficacy of the Project ÒRÉ intervention.
Conduct a qualitative process evaluation | 18 Months
  To conduct a qualitative process evaluation to assess the acceptability of the experimental intervention in a new community using a subset of the participants in the experimental condition.

CONTACTS AND LOCATIONS:
Overall Officials: M. Margaret Dolcini, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States